CLINICAL TRIAL: NCT04594330
Title: Pilot Trial for the Benefit of Virgin Coconut Oil (VCO) as a Potential Adjuvant Therapy in COVID-19 Patients
Brief Title: Virgin Coconut Oil (VCO) as a Potential Adjuvant Therapy in COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Ika Trisnawati, dr., MSc., internist-pulmonologist, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002/05/2020
Record Dates: First submitted 2020-10-05; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Infections
Keywords: COVID-19; treatment; virgin coconut oil
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Mineral Waters

STUDY DESIGN:
Intervention Model Description: The COVID-19 patients are recruited according to the inclusion and exclusion criteria, then divided into two groups. Group I, the intervention group, consists of COVID-19 patients receiving standard therapy and 15 mL of VCO twice a day for 14 days. Group II, the control group, consists of COVID-19 patients receiving standard therapy and 15 mL of placebo twice a day for 14 days.
Who Masked: Participant, Care Provider
Masking Description: The participants and care provider are blinded to the type of treatment that the participants receive.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - 30 COVID-19 patients aged ≥ 18 years old receiving the investigational drug (Active Comparator): Group 1 - 30 COVID-19 patients receiving standard therapy and the investigational drug (Virgin Coconut Oil)
  Interventions: Drug: virgin coconut oil (VCO)
- Group 2 - 30 COVID-19 patients aged ≥ 18 years old receiving placebo (Placebo Comparator): Group 2 - 30 COVID-19 patients receiving standard therapy and placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: virgin coconut oil (VCO) — 15 mL of VCO twice a day for 14 days
  Other Names: virgin coconut oil
  Arms: Group 1 - 30 COVID-19 patients aged ≥ 18 years old receiving the investigational drug
Other: placebo — 15 mL of placebo twice a day for 14 days
  Other Names: mineral water
  Arms: Group 2 - 30 COVID-19 patients aged ≥ 18 years old receiving placebo

SUMMARY:
Virgin Coconut Oil (VCO) contains multiple compounds which have antibacterial, antiviral, and immunomodulatory properties. The role of VCO as an antivirus to treat COVID-19 requires further studies. A previous study has investigated the used of 30 ml of VCO to healthy volunteers for a month and reported no side effect. Here the investigators conduct a pilot trial to investigate the effect of VCO towards the clinical outcomes of COVID-19 patients in Indonesia.

DETAILED DESCRIPTION:
The subjects of this pilot study are patients diagnosed with COVID-19 in Central Public Hospital Dr. Sardjito, Teaching Hospital of Universitas Gadjah Mada (UGM), and Yogyakarta COVID-19 referral hospitals (RSUD Wonosari and Sleman). The COVID-19 patients are recruited according to the inclusion and exclusion criteria, then divided randomly into two groups. Group I, the intervention group, consists of COVID-19 patients receiving standard therapy and 15 mL of VCO twice a day for 14 days. Group II, the control group, consists of COVID-19 patients receiving standard therapy and 15 mL of placebo twice a day for 14 days. Both groups are monitored for four weeks with a nasopharyngeal or oropharyngeal Polymerase Chain Reaction (PCR) swab test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥ 18 years old.
* COVID-19 patients diagnosed with nasopharyngeal/oropharyngeal PCR swab specimens that are treated in Central Public Hospital Dr. Sardjito, Teaching Hospital of Universitas Gadjah Mada (UGM), and Yogyakarta COVID-19 referral hospitals.
* Patients with mild and moderate pneumonia symptoms that are treated in Central Public Hospital Dr. Sardjito, Teaching Hospital of Universitas Gadjah Mada (UGM), and Yogyakarta COVID-19 referral hospitals.

Exclusion Criteria:

* Patients with liver function disorder.
* VCO hypersensitivity.
* Patients with severe pneumonia and/or Acute Respiratory Distress Syndrome (ARDS).
* Pregnant patients.
* Patients with malignant comorbidity.
* Critical or unconscious patients.
* Patients using other immunomodulators similar to VCO within less than three days before VCO administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Ordinal scale for measuring clinical improvement by the World Health Organization (WHO) | 14 days
  Clinical improvement determined by the World Health Organization (WHO) in ordinal scale (0-8)
Clinical symptoms improvement, determined with interview and examination | 14 days
  Duration of symptoms (fever, respiratory rate or shortness of breath, and cough) that is calculated according to the start of VCO or placebo administration until symptoms disappear, obtained based on anamnesis and physical examination
Pain as side effects of the drugs, measured by Visual Analog Scale | 14 days
  Probable side effects of the virgin coconut oil, i.e. headache, stomachache, muscle pain, measured in Visual Analog Scale (0-10)
Allergic reaction severity in mild, moderate, or severe | 14 days
  Probable side effects of the virgin coconut oil, i.e. allergic reaction severity, categorized in mild, moderate, or severe reaction.

SECONDARY OUTCOMES:
Laboratory outcome of leucocyte count | 14 days
  leucocyte count, measured in 1000/micro liter
Laboratory outcome of lymphocyte count | 14 days
  lymphocyte count, measured in percentage
Laboratory outcome of neutrophil count | 14 days
  Neutrophil count, measured in percentage
Laboratory outcome of neutrophil to lymphocyte ratio, in scale | 14 days
  neutrophil to lymphocyte ratio, in scale
Laboratory outcome of D-dimer | 14 days
  D-dimer measured in microgram/Liter
Laboratory outcome of TNF-alpha | 14 days
  TNF-alpha, measured in pg/ml
Laboratory outcome of CRP value | 14 days
  CRP value measured in qualitative value
Laboratory outcome of IL-6 | 14 days
  IL-6 value measured in pg/ml
Laboratory outcome of ferritin | 14 days
  Ferritin value measured in mcg/liter
Laboratory outcome of procalcitonin | 14 days
  procalcitonin in microgram/liter
chest radiology outcome, measured as improvement of infiltrate based on expert assessment | 14 days
  chest radiology outcome, measured as improvement of infiltrate based on expert assessment in day 1 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Ika Trisnawati, MD, MSc, internist, Principal Investigator — Gadjah Mada University
Locations (4):
- Indonesia (4):
  - Central Public Hospital Dr. Sardjito, Yogyakarta
  - RSUD Wonosari, Yogyakarta
  - RSUP Sleman, Yogyakarta
  - Teaching Hospital of Universitas Gadjah Mada (UGM), Yogyakarta

IPD SHARING:
Plan to Share IPD: No